CLINICAL TRIAL: NCT00414739
Title: Testing of Innocuousness of Benzalkonium Chloride on the Eye Concerning Possible Growth of Langerhans Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BAC-2006-1
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Eye Diseases
Keywords: growth of dendritic cells; prevention
MeSH Terms: conditions — Eye Diseases | interventions — Benzalkonium Compounds

INTERVENTIONS:
Drug: Benzalkonium chloride

SUMMARY:
The study analysis the influence of benzalkonium chloride on the density of antigen presenting Langerhans cells. This is achieved in a double blind randomized study using in-vivo confocal microscopy to identify and quantify Langerhans cells of the human cornea in its central and peripheral part. This study design is based on observations with raised Langerhans cell density after the application of benzalkonium chloride containing eye drops in glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy probands

Exclusion Criteria:

* eye diseases
* pregnancy and lactation period
* drug dependency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20

PRIMARY OUTCOMES:
Possible raised Langerhans cell density in the corneal epithelium

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf F. Guthoff, Prof. Dr., Study Chair — University of Rostock, Eye Department
Locations (1):
- University of Rostock, Eye Department, Rostock, Germany

REFERENCES:
- [Background] De Saint Jean M, Brignole F, Bringuier AF, Bauchet A, Feldmann G, Baudouin C. Effects of benzalkonium chloride on growth and survival of Chang conjunctival cells. Invest Ophthalmol Vis Sci. 1999 Mar;40(3):619-30. PMID 10067965
- [Background] Becquet F, Goldschild M, Moldovan MS, Ettaiche M, Gastaud P, Baudouin C. Histopathological effects of topical ophthalmic preservatives on rat corneoconjunctival surface. Curr Eye Res. 1998 Apr;17(4):419-25. doi: 10.1080/02713689808951223. PMID 9561834
- [Background] Noecker R. Effects of common ophthalmic preservatives on ocular health. Adv Ther. 2001 Sep-Oct;18(5):205-15. doi: 10.1007/BF02853166. PMID 11783457
- [Background] Eckard A, Stave J, Guthoff RF. In vivo investigations of the corneal epithelium with the confocal Rostock Laser Scanning Microscope (RLSM). Cornea. 2006 Feb;25(2):127-31. doi: 10.1097/01.ico.0000170694.90455.f7. PMID 16371768
- [Background] Zhivov A, Stachs O, Kraak R, Stave J, Guthoff RF. In vivo confocal microscopy of the ocular surface. Ocul Surf. 2006 Apr;4(2):81-93. doi: 10.1016/s1542-0124(12)70030-7. PMID 16681079
- [Background] Zhivov A, Stave J, Vollmar B, Guthoff R. In vivo confocal microscopic evaluation of Langerhans cell density and distribution in the normal human corneal epithelium. Graefes Arch Clin Exp Ophthalmol. 2005 Oct;243(10):1056-61. doi: 10.1007/s00417-004-1075-8. Epub 2005 Oct 20. PMID 15856272